CLINICAL TRIAL: NCT00168506
Title: Panic Disorder and Cardiac Risk: Evaluation of a Psychological Treatment Which Addresses Biology, Psychology and Behaviour
Brief Title: Panic Disorder and Cardiac Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baker Heart Research Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHMRC P - 01
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Panic Disorder
Keywords: panic disorder; cardiac risk
MeSH Terms: conditions — Panic Disorder

INTERVENTIONS:
Drug: SSRI
Drug: CBT
Drug: CBT/SSRI

SUMMARY:
The reason for increased cardiac mortality in panic disorder has not been precisely identified, but possibly is due to chronic activation of the cardiac stimulant (sympathetic) nerves, which may predispose the individual with panic disorder to disorders of cardiac rhythm and coronary artery spasm. The uniqueness of this study lies in its comprehensive evaluation of a psychobiological approach to the treatment of panic disorder using change in biological, behavioural and psychological variables as criteria for efficacy. 50 patients aged between 18 and 60 years will be recruited; both males and females. They will be treated with either cognitive behavioural therapy (CBT) or SSRI (selective serotonin re-uptake inhibitor) antidepressants or a combination of both.

This project will firstly compare individuals with panic disorder who demonstrate abnormal brain transmitter (noradrenaline, serotonin) with those who demonstrate normal activity of these neurotransmitters, on interoceptive accuracy for changes in sympathetic nervous system arousal. It is predicted that individuals who demonstrate abnormal activity of these neurotransmitters will also demonstrate enhanced interoceptive ability to detect changes in arousal levels. Secondly, this project will evaluate the effects of a psychobiological treatment approach to panic disorder involving a combination of CBT and SSRI. This approach will be compared to the effects of both these interventions alone on a comprehensive array of measures related to panic disorder. It is predicted that the combined approach will be the most effective intervention on behavioural, psychological and biological variables, and cardiac risk. We will also be able to assess whether changes in panic disorder severity are associated with changes in interoceptive accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Panic disorder

Exclusion Criteria:

* Comorbid heart disease
* Comorbid significant psychiatric illness
* Significant suicide risk
* HIV/AIDS hepatitis B/c

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-06; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Murray A Esler, MBBS Phd, Principal Investigator — Baker Heart Research Insitute
Locations (1):
- Baker Heart Research Institute, Melbourne, Victoria, Australia